CLINICAL TRIAL: NCT06006091
Title: Clinical Outcomes of Letrozole-induced Endometrial Preparation Regimens Versus Conventional Endometrial Preparation Regimens Including Natural Cycle, Hormone Replacement Regimens in FET, a Randomized Controlled Study
Brief Title: The Effectiveness of the Letrozole-induced Endometrial Preparation Protocol in Frozen-thawed Embryo Transfer (FET)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Chenliang Zhou, Director, International Peace Maternity and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: InternationalPMCHH-1
Record Dates: First submitted 2023-07-31; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Letrozole; Infertility, Female
Keywords: Frozen-thawed embryo transfer; Letroziole; Endothelial preparation protocol
MeSH Terms: conditions — Infertility, Female | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Letrozole-induced endometrial preparation protocol (Experimental): Starting at D3 of the menstrual cycle, letrozole 2.5 mg po qd was administered for 5 days. After 1 week, ultrasound was performed to dynamically monitor follicular development, and 75-150 IU im qd of human menopausal gonadotrophin (hMG) given to continue ovulation stimulation as needed, and oestradiol valerate 2 mg po qd was given to regulate endometrial thickness until the follicle developed to 16 mm in diameter and 7 mm in endometrial thickness. The follicles developed to ≥16 mm in diameter and ≥7 mm in lining thickness and were dynamically monitored by ultrasound and serum sex hormone levels to determine the day of ovulation. From the day of ovulation, dexamethasone 10 mg po tid was administered, and cleavage-stage embryos were transferred 2 or 3 days later, or blastocysts were transferred 5 days later. Deferiprone 10 mg po tid was continued for 14 days after transfer.
  Interventions: Drug: Letrozole
- Natural cycles endometrial preparation protocol (No Intervention): Follicular development was monitored dynamically by ultrasound from D8-D11of the menstrual cycle until the follicles developed to ≥16 mm in diameter and ≥7 mm in endothelial thickness, and the day of ovulation was determined by dynamic ultrasound monitoring and detection of serum sex hormone levels. Deferiprone 10 mg po tid was administered from the day of ovulation, and D2 or D3 cleavage stage embryos were transferred 2 or 3 days later, or blastocysts were transferred 5 days later. Deferiprone 10 mg po tid was continued for a total of 14 days after transfer. Cycles were canceled if endothelial thickness was <7 mm on the day of ovulation or if serum progesterone levels were 5 nmol/L before ovulation.
- Hormone replacement cycles endometrial preparation protocol (No Intervention): Starting from D1-D5 of the menstrual cycle, estradiol valerate 2 mg po bid was administered for 7 days, followed by ultrasound for dynamic monitoring of endothelial and follicular development, and if the endothelial thickness was <7 mm, the dosage of estradiol valerate was increased to 3-4 mg po bid as appropriate. The number of days of hormone replacement ranged from 11-20 days, and when the endothelial thickness was 7 mm, luteinizing hormone vaginal slow-release gel 90 mg pv qd was added, as well as dexedrine and progesterone 10 mg po bid to transform the endothelium 2 or 3 days later or 5 days later. Progesterone 10 mg po bid was added to transform the endothelium, and cleavage stage embryos were transferred 2 or 3 days later, or blastocysts were transferred 5 days later. Luteal support as described above was continued for a total of 14 days after transfer.

INTERVENTIONS:
Drug: Letrozole — Different endothelial preparations according to groups, see arm descriptions for details
  Arms: Letrozole-induced endometrial preparation protocol

SUMMARY:
The goal of this single center, non-blinded, randomized controlled clinical trial to comparison of pregnancy outcomes and perinatal outcomes in patients undergoing IVF treatment (including ICSI) with FET with letrozole-induce endothelial preparation protocol versus natural cycles, hormone replacement protocol.

The main questions it aims to answer are:

* To investigate whether letrozole-induce endothelial preparation is effective in improving the live birth rate and clinical pregnancy rate.
* To explore its possible impact on clinically important indicators such as spontaneous abortion rate, implantation cycle cancellation rate, days of endothelial preparation, and number of visits to the clinic.

The study subjects were randomized into groups starting at D1-D3 of the menstrual cycle. The study subjects were stratified according to whether their menstrual cycles were regular or not, and were divided into the following endothelial preparation regimens according to the pre-prepared stratified zoned randomized group numbers: (1) regular menstrual cycles (25-35 d): letrozole ovulation-promoting cycles, natural cycles, and hormone-replacement cycles; and (2) irregular menstrual cycles (<25 d or >35 d): letrozole ovulation-promoting cycles, hormone-replacement cycle.

ELIGIBILITY:
Inclusion Criteria:

Women <40 years of age undergoing IVF or ICSI at our reproductive center with a total of ≤3 superovulation cycles , and with ≥2 cleavage embryos or ≥1 blastocyst were cryopreserved. Previous cycles of embryo transfer ≤ 2 and only one transfer cycle with 1-2 embryos per study subject was enrolled.

Exclusion Criteria:

1. Patients with chromosomal abnormalities in either spouse, hydrosalpinx, severe endometriosis, adenomyosis, and uterine and uterine cavity organic diseases such as uterine malformations, endometrial polyps, and uterine adhesions;
2. patients who underwent pre-implantation genetic diagnosis (PGT);
3. patients who underwent ICSI using surgically obtained epididymal or testicular spermatozoa;
4. patients with a Body mass index (BMI, = weight/height2 ) > 30 kg/m2;
5. patients with recurrent spontaneous abortions;
6. patients with sequential embryo transfer.

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — As this was an assisted reproduction-related study, the population included was physiologically (with uterus and ovaries) and genetically (with XX sex chromosomes) female.
Enrollment: 858 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Live birth | 40-42 weeks'estimated gestational age
  The number of deliveries resulting in at least one live birth

SECONDARY OUTCOMES:
Clinical pregnancy | 5-7 weeks' estimated gestational age
  Clinical pregnancies diagnosed by ultrasonographic visualisation of gestational sacs, the number of clinical pregnancies expressed per 100 embryo transfer cycles
embryo implantation | 14 day after embryo transfer
  Serum Human Chorionic Gonadotropin levels >10 IU/L, the number of gestational sacs observed divided by the number of embryos transferred

CONTACTS AND LOCATIONS:
Locations (1):
- Yu Xiao, Shanghai, China